CLINICAL TRIAL: NCT01677247
Title: Bioequivalence Study of Two Formulations of Glimepiride Tablet in Healthy Subjects
Brief Title: Bioequivalence Study of 4 mg Glimepiride Tablet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BE-Glimepiride
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Glimepiride BE Study in Healthy Volunteers Under Fasting Condition
Keywords: sulphonylurea; anti-hyperglycaemic; bioavailability; bioequivalence; glimepiride; pharmacokinetics
MeSH Terms: interventions — glimepiride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I (Test) (Experimental): Test : glimepiride 4 mg tablet of PT Dexa Medica
  Interventions: Drug: Group I (Test) : Glimepiride 4 mg tablet of PT Dexa Medica
- Group II (Reference) (Active Comparator): Reference : glimepiride (Amaryl) 4 mg tablet of PT Sanofi-Aventis, Indonesia
  Interventions: Drug: Group II (Reference) : glimepiride (Amaryl) 4 mg tablet of PT Sanofi Aventis

INTERVENTIONS:
Drug: Group I (Test) : Glimepiride 4 mg tablet of PT Dexa Medica — In each of the two study periods (separated by a washout of one week) a single dose of test or reference product was administered.
  Arms: Group I (Test)
Drug: Group II (Reference) : glimepiride (Amaryl) 4 mg tablet of PT Sanofi Aventis — In each of the two study periods (separated by a washout of one week) a single dose of test or reference product was administered.
  Other Names: Amaryl®, manufactured by PT Sanofi Aventis
  Arms: Group II (Reference)

SUMMARY:
This was a randomized, single blind, two-period, two sequence cross-over study under fasting condition to compare the bioavailability of two glimepiride 4 mg tablet formulations (test and reference formulations).

DETAILED DESCRIPTION:
The participating subjects were required to have an overnight fast; and in the next morning they were given orally either one tablet of 4 mg glimepiride as the test drug (produced by PT Dexa Medica) or one tablet of 4 mg glimepiride (Amaryl®, Sanofi Aventis) as the reference drug with 200 mL water.

Blood samples were drawn immediately before taking the drug (control), and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4.5, 6, 9, 12, 18 and 24 hours after drug administration. Immediately after drug administration, subjects were administered 100 ml of 10% glucose at approximately 0.5, 1.5, 2, 2.5, 3.5, and 4.5 hours. In addition, 20% glucose solution was given to any subject who exhibited symptoms of hypoglycaemia. One week after the first drug administration (wash-out period), the procedure was repeated using the alternate drug.

The plasma concentrations of glimepiride were determined by high performance liquid chromatography with ultraviolet detection (HPLC-UV). The pharmacokinetic parameters assessed are AUCt, AUCinf, Cmax, tmax, and t1/2.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects with absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluation, medical history or physical examination during screening
2. Age of 18 - 55 years
3. Preferably non-smokers or moderate smokers (less than 10 cigarettes per day)
4. Able to participate, communicate well with the investigators and willing to provide written informed consent to participate in the study
5. BMI 18 - 25 kg/m2
6. Vital signs (after 10 minutes rest) must be within the following ranges:

   * SBP 100 - 120 mmHg
   * DBP 60 - 80 mmHg
   * Pulse rate 60 - 90 bpm

Exclusion Criteria:

1. Personal/family history of allergy or hypersensitivity or contraindication to glimepiride or allied drugs
2. Pregnant or lactating women
3. Any major illnesses in the past 90 days or clinically significant ongoing chronic medical illness
4. Presence of any clinically significant abnormal values during screening
5. Positive Hepatitis B surface antigen (HBsAg), anti-HCV, or anti-HIV
6. Clinically significant haematology abnormalities
7. Clinically significant electrocardiogram (ECG) abnormalities
8. Any surgical or medical condition (present or history) which might significantly alter the absorption, distribution, metabolism or excretion of the study drug
9. Past history of anaphylaxis or angioedema
10. History of drug or alcohol abuse within 12 months prior to screening
11. Participation in any clinical trial within the past 90 days
12. History of any bleeding or coagulative disorders
13. History of difficulty with donating blood or difficulty in accessibility of veins in left or right arm
14. A donation or loss of 500 mL (or more) of blood within 3 months before this study's first dosing day
15. Intake of any prescription, non-prescription drug, food supplements or herbal medicines within 14 days of this study's first dosing day

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Bioavailability | 24 hours
  Relative bioavailability (primarily measured by AUC and Cmax) between two glimepiride 4 mg tablet formulations (test and reference formulations) under fasting condition.

SECONDARY OUTCOMES:
Bioavailability | 24 hours
  Relative bioavailability (secondarily measured by tmax and t1/2) between two formulations of glimepiride 4 mg tablets (the Test and Reference formulations)
Adverse events | 1 months
  The presence of adverse events will be observed, reported and sufficiently handled during subjects' participation in the study (1 month).

CONTACTS AND LOCATIONS:
Overall Officials: Danang A. Yunaidi, MD, Principal Investigator — PT Equilab International
Locations (1):
- PT Equilab International, Jakarta, Jakarta Special Capital Region, Indonesia

REFERENCES:
- [Background] Salem II, Idrees J, Al Tamimi JI. Determination of glimepiride in human plasma by liquid chromatography-electrospray ionization tandem mass spectrometry. J Chromatogr B Analyt Technol Biomed Life Sci. 2004 Jan 5;799(1):103-9. doi: 10.1016/j.jchromb.2003.10.024. PMID 14659441
- [Background] Jovanovic D, Stojsic D, Zlatkovic M, Jovic-Stosic J, Jovanovic M. Bioequivalence assessment of the two brands of glimepiride tablets. Vojnosanit Pregl. 2006 Dec;63(12):1015-20. doi: 10.2298/vsp0612015j. PMID 17252706
- [Background] Malerczyk V, Badian M, Korn A, Lehr KH, Waldhausl W. Dose linearity assessment of glimepiride (Amaryl) tablets in healthy volunteers. Drug Metabol Drug Interact. 1994;11(4):341-57. doi: 10.1515/dmdi.1994.11.4.341. PMID 12369757